CLINICAL TRIAL: NCT01817686
Title: Default Options in Advance Directives for Veterans With Serious Illnesses: A Randomized Clinical Trial
Brief Title: Study of Default Options in Advance Directives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua B. Kayser, Assistant Professor of Clinical Medicine, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01381
Record Dates: First submitted 2013-03-19; First posted 2013-03-25 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: COPD; Severe or Very Severe Airflow Obstruction and/or Receiving or Eligible to Receive Long-term Oxygen Therapy; Idiopathic Pulmonary Fibrosis; Other Interstitial Lung Disease Without Curative Therapy; Congestive Heart Failure; NYHA Class IV or NYHA Class III Plus 1 Hospitalization in the Past Year; Malignancy; Any Stage 3B or 4 Solid Tumor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis; Heart Failure; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Comfort Default (Experimental): ADs with pre-selected defaults that focus on providing comfort at end-of-life.
  Interventions: Other: Comfort Default AD forms
- Life Extension Default (Experimental): ADs with pre-selected defaults that focus on extending life.
  Interventions: Other: Life Extension Default AD forms
- Standard Default (Experimental): ADs without pre-selected defaults.
  Interventions: Other: Standard Default AD forms

INTERVENTIONS:
Other: Comfort Default AD forms — Consenting subjects will be randomly assigned to one of 3 study arms. Subjects will receive a different AD form based on which arm they have been randomly assigned. Once a completed AD form is received, a debriefing session will be held to alert patients to exactly how the 3 ADs used in the study differ. Once patients are fully informed about the variations in the ADs, the patients will have an opportunity to change their AD selections prior to finalizing them as a part of their medical record. A final satisfaction interview will take place with a research associate who will contact patients via telephone to administer a satisfaction questionnaire.
  Arms: Comfort Default
Other: Life Extension Default AD forms — Consenting subjects will be randomly assigned to one of 3 study arms. Subjects will receive a different AD form based on which arm they have been randomly assigned. Once a completed AD form is received, a debriefing session will be held to alert patients to exactly how the 3 ADs used in the study differ. Once patients are fully informed about the variations in the ADs, the patients will have an opportunity to change their AD selections prior to finalizing them as a part of their medical record. A final satisfaction interview will take place with a research associate who will contact patients via telephone to administer a satisfaction questionnaire.
  Arms: Life Extension Default
Other: Standard Default AD forms — Consenting subjects will be randomly assigned to one of 3 study arms. Subjects will receive a different AD form based on which arm they have been randomly assigned. Once a completed AD form is received, a debriefing session will be held to alert patients to exactly how the 3 ADs used in the study differ. Once patients are fully informed about the variations in the ADs, the patients will have an opportunity to change their AD selections prior to finalizing them as a part of their medical record. A final satisfaction interview will take place with a research associate who will contact patients via telephone to administer a satisfaction questionnaire.
  Arms: Standard Default

SUMMARY:
Default options represent the events or conditions that are set into place if no alternatives are actively chosen. The setting of default options has well-established effects on a broad range of human decisions, but its influence on patients' preferences for end-of-life care is only beginning to be understood.

This is a 3-armed randomized clinical trial in Veterans at high risk for critical illness, assessing the impact of Advance Directive (AD) forms framed with different default options. The central goals are to assess how default options in ADs influence the end-of-life care choices made by patients at risk for critical care, and these patients' hospital and ICU utilization.

The investigators hypothesize that setting defaults in real ADs will increase the proportion of Veterans selecting comfort-oriented plans of care, decrease selections of life-extending therapies such as mechanical ventilation and dialysis, and reduce the proportion of time during follow-up that Veterans spend in the hospital and/or ICU, without affecting patient satisfaction with end-of-life care planning.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Chronic Obstructive Pulmonary Disease (COPD) with severe or very severe airflow obstruction on pulmonary function testing and or receiving or eligible to receive long-term oxygen therapy AND/OR
* Idiopathic Pulmonary Fibrosis (IPF) AND/OR
* Other interstitial lung disease without curative therapy AND/OR
* Any stage 3B or 4 solid tumor AND/OR
* Congestive Heart Failure (CHF) either New York Heart Association NYHA) class IV or NYHA class III plus 1 hospitalization in the past year
* No previously signed advance directive in the medical record
* Neither listed for nor considering lung or heart transplantation
* High anticipated risk for critical illness in the next 2 years based on clinical judgment
* Interest in thinking about filling out an Advance Directive

Exclusion Criteria:

* Diseases for which life-extending medical therapies may be available
* Inability to speak and/or read English proficiently
* New clinic patients meeting the clinic provider for the first time
* Patients being actively evaluated or already listed for transplants
* Patients already having an AD
* Cognitive impairment necessitating proxy consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evaluate how the setting of defaults influences the proportion of Veterans selecting comfort-oriented plans of care in real ADs | 18 months
  The primary outcome is the proportion of patients in each of the 3 groups who select a general plan of care that prioritizes comfort over life extension.

SECONDARY OUTCOMES:
Assess the influence of default options in ADs on Veterans' selections of specific life-extending therapies | 18 months
  The proportions of patients electing to receive each of the 5 specific life-extending interventions
Determine whether setting defaults in ADs influences the proportion of time during follow-up that Veterans spend in the hospital or ICU | 18 months
  The proportion of time during a 6-18 month follow-up (median 1 year) that patients spend in the hospital or ICU for each AD group

OTHER OUTCOMES:
To document feasibility of a study of Advance Directives in the Veteran population | 18 months
  To document our ability to recruit and retain patients with advanced diseases, we will measure the proportions of patients approached for consent who enroll (consent rate), the proportion of such patients who complete their AD (completion rate), and the proportion who subsequently complete their advance care satisfaction interview (retention rate).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua B Kayser, MD, MPH, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania, United States